CLINICAL TRIAL: NCT06742112
Title: Validity and Reliability of the 6-minute Pegboard and Ring Test in Assessing Upper Extremity Function in Overweight and Obese Individuals
Brief Title: The 6-minute Pegboard and Ring Test in Overweight and Obese Individuals
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2024-20/173
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Overweight or Obese Adults
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Overweight and obese individuals

SUMMARY:
The aim of our study is to investigate the validity and reliability of the 6-minute pegboard and ring test in overweight and obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 25 kg/m2
* Volunteering for the study

Exclusion Criteria:

* Having uncontrolled hypertension, diabetes mellitus
* Having comorbidities that may affect physical functions
* Failure to cooperate with tests to be performed
* Liver disease, kidney disease, cancer, lung diseases and serious cardiomyopathies, neurological diseases
* Pregnancy
* Having a history of bariatric surgery
* Presence of contraindications to exercise testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overweight and obese individuals will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Arm exercise capacity | 1st day
  It will be assessed by 6 minute pegboard and ring test.
Exercise capacity | 1st day
  It will be assessed by 6 minute walk test.
Hand grip strength | 1st day
  Will be measured using a hang grip dynamometer.
Muscle endurance | 1st day
  30 second push-up test will be used, and total number will be recorded.

SECONDARY OUTCOMES:
Upper extremity functional status | 1st day
  Upper extremity functional status will be assessed with the Upper Extremity Functional Index. This index consists of 20 questions, and the lowest possible score is 0 and the highest score is 80. Higher scores indicate better functional status.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided